CLINICAL TRIAL: NCT00547196
Title: Allogeneic Stem Cell Transplantation for Patients With Hematological Malignancies Using Multiple Unrelated Cord Blood Units
Brief Title: AlloHCT From Matched Unrelated Donors in Pts w/ Advanced Hematologic Malignancies & Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02165; P30CA033572 (NIH); CHNMC-02165; CDR0000570249 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2023-04-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: refractory chronic lymphocytic leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute lymphoblastic leukemia in remission; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; relapsing chronic myelogenous leukemia; recurrent cutaneous T-cell non-Hodgkin lymphoma; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Cutaneous | interventions — Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Melphalan; Mycophenolic Acid; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen I (FTBI, Cyclophosphamide, Fludarabine) (Experimental): Patients undergo FTBI 2-3 times a day on days -9 to -6 for a total of 11 fractions. Patients also receive cyclophosphamide IV over 2 hours on days -5 and -4 and fludarabine phosphate IV on days -5 to -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  Interventions: Biological: filgrastim; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine phosphate; Drug: Mycophenolate Mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: umbilical cord blood transplantation; Radiation: Fractionated total body irradiation
- Regimen II (Busulfan, Fludarabine, Melphalan) (Experimental): Patients receive a test dose of busulfan on day -10 and then dose adjusted busulfan IV 3-4 times daily on days -9 to -6, melphalan IV on days -5 and -4, and fludarabine phosphate IV on days -5 to -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  Interventions: Biological: filgrastim; Drug: Busulfan; Drug: Cyclosporine; Drug: Fludarabine phosphate; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: umbilical cord blood transplantation
- Regimen III (TBI, Cyclophosphamide, Fludarabine) (Experimental): Patients receive fludarabine phosphate IV on days -8 to -4 and cyclophosphamide IV over 2 hours on day -3 and undergo TBI (single dose) on day -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  Interventions: Biological: filgrastim; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine phosphate; Drug: Mycophenolate Mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: umbilical cord blood transplantation; Radiation: total-body irradiation
- Regimen IV (Fludarabine, Melphalan) (Experimental): Patients receive fludarabine phosphate IV on days -7 to -3 and melphalan IV on day -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  Interventions: Biological: filgrastim; Drug: Cyclosporine; Drug: Fludarabine phosphate; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: Busulfan
  Other Names: Busilvex
  Arms: Regimen II (Busulfan, Fludarabine, Melphalan)
Drug: Cyclophosphamide
  Other Names: CTX
  Arms: Regimen I (FTBI, Cyclophosphamide, Fludarabine); Regimen III (TBI, Cyclophosphamide, Fludarabine)
Drug: Cyclosporine
  Other Names: CsA
Drug: Fludarabine phosphate
  Other Names: Fludara
Drug: Melphalan
  Other Names: Alkeran
  Arms: Regimen II (Busulfan, Fludarabine, Melphalan); Regimen IV (Fludarabine, Melphalan)
Drug: Mycophenolate Mofetil
  Other Names: MMF
Procedure: allogeneic hematopoietic stem cell transplantation
  Other Names: AlloHCT
Procedure: umbilical cord blood transplantation
Radiation: total-body irradiation
  Other Names: TBI
  Arms: Regimen III (TBI, Cyclophosphamide, Fludarabine)
Radiation: Fractionated total body irradiation
  Other Names: FTBI
  Arms: Regimen I (FTBI, Cyclophosphamide, Fludarabine)

SUMMARY:
RATIONALE: Giving chemotherapy with or without total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil before and after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well four different chemotherapy regimens given with or without total-body irradiation before umbilical cord blood transplant work in treating patients with relapsed or refractory hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the survival at day 100 of patients with relapsed, refractory, or poor-risk hematological malignancies treated with four different preparative regimens followed by allogeneic hematopoietic stem cell transplantation (HSCT) using two unrelated umbilical cord blood (UCB) units.

Secondary

* To determine the incidence and timing of neutrophil engraftment in patients treated with these regimens.
* To determine the incidence and timing of platelet engraftment in patients treated with these regimens.
* To determine the incidence and severity of acute and chronic graft-versus-host-disease (GVHD) in patients treated with these regimens.
* To determine the survival at day 180 in patients treated with these regimens.
* To determine the disease-free survival in patients treated with these regimens.
* To determine the incidence of primary and secondary engraftment failure in patients treated with these regimens.
* To determine the incidence of transplantation-related complications (e.g., infection, veno-occlusive disease of the liver, or organ toxicity) in these patients.
* To determine the incidence of post-transplantation-related lymphoproliferative disease, secondary myelodysplastic syndromes, or other secondary malignancies in these patients.
* To determine the incidence of relapse in patients treated with these regimens.
* To determine post-transplantation chimerism in patients treated with these regimens.
* To determine immune reconstitution in patients treated with these regimens.

OUTLINE: This is a multicenter study.

* Preparative regimens: Patients are assigned to 1 of 4 preparative regimens.

  * Regimen 1 (for patients < 50 years of age and no contraindication to fractionated total-body irradiation (FTBI): Patients undergo FTBI 2-3 times a day on days -9 to -6 for a total of 11 fractions. Patients also receive cyclophosphamide IV over 2 hours on days -5 and -4 and fludarabine phosphate IV on days -5 to -2.
  * Regimen 2 (for patients < 50 years of age and unable to tolerate FTBI due to prior dose-limiting radiotherapy or significant cardiotoxicity): Patients receive a test dose of busulfan on day -10 and then dose adjusted busulfan IV 3-4 times daily on days -9 to -6, melphalan IV on days -5 and -4, and fludarabine phosphate IV on days -5 to -2.
  * Regimen 3* (for patients unable to tolerate regimen 1 or 2; no age exclusion): Patients receive fludarabine phosphate IV on days -8 to -4 and cyclophosphamide IV over 2 hours on day -3 and undergo TBI (single dose) on day -2.
  * Regimen 4* (for patients unable to tolerate regimen 1 or 2): Patients receive fludarabine phosphate IV on days -7 to -3 and melphalan IV on day -2.

NOTE: *Treating physician decides the choice between regimen 3 and 4

* Umbilical cord blood (UCB) transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover.
* Graft-versus-host-disease prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hematological or lymphatic malignancy, including any of the following:

  * Acute myeloid leukemia

    * Relapsed or primary refractory disease with < 10% blasts on peripheral blood smear
    * In first remission with poor risk factors and molecular prognosis [i.e., AML with -5, -7, t(6;9), tri8, -11] (preparative regimen 3 or 4)
  * Acute lymphocytic leukemia

    * In second complete remission or higher OR in first remission with poor risk factors, including any of the following (preparative regimen 1 or 2):

      * BCR/ABL by fluorescence in situ hybridization (FISH) or reverse transcriptase-polymerase chain reaction
      * t(9;22)(q34;q11) detected by cytogenetics
      * Chromosomes < 44 by cytogenetics
      * DNA index < 0.81 by flow cytometry
      * Any rearrangement of chromosome 11 that results in disruption of MLL gene (11q23) by cytogenetics and SER
    * In first remission with poor risk factors and molecular prognosis [ALL with Philadelphia chromosome-positive t(9;22), t(4;22), (q34;q11)] (preparative regimen 3 or 4)
  * Chronic myelogenous leukemia

    * In accelerated phase or greater (preparative regimen 1 or 2)
    * In accelerated or second chronic phase (preparative regimen 3 or 4)
  * Myelodysplastic syndromes

    * With deletion of chromosome 7 or short arm of chromosome 5 (preparative regimen 1 or 2)
    * In high and high-intermediate risk categories (preparative regimen 3 or 4)
  * Non-Hodgkin lymphoma in relapse with marrow involvement
  * Refractory chronic lymphocytic leukemia
* Patients deemed ineligible for conventional high-dose chemotherapy programs (i.e., regimens 1 or 2) due to any of the following concurrent medical conditions may be eligible for regimens 3 or 4 at the discretion of the treating physician and principal investigator (preparative regimen 3 or 4):

  * LVEF < 50% and > 40%
  * FEV1, FVC, or DLCO < 50%
  * Bilirubin > 3 mg/dL
  * Creatinine > 2 mg/dL
* Two partially HLA-matched umbilical cord blood (UCB) units available

  * HLA-matched minimally at 4 of 6 HLA-A, HLA-B, and -DRB1 loci with the patient

    * DRB1 matched by high resolution DNA typing
    * HLA-A and HLA-B matched by low resolution at the "serological match" level
  * Two pooled units with a nucleated cell number > 2.5 x 10^7/kg
* No available HLA-identical sibling or 1 antigen-mismatched related donor
* No available HLA-matched unrelated bone marrow donor

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* Karnofsky performance status (PS) 60-100% OR Lansky PS 60-100% OR Zubrod PS 0-1
* Physiological age 60 or less (at any chronological age)
* Weight > 50 kg
* Creatinine normal for age OR creatinine clearance by 24-hour urine collection or glomerular filtration rate > 60 mL/min
* Bilirubin ≤ 1.5 mg/dL
* LVEF ≥ 50%
* DLCO ≥ 60% of predicted
* No HIV-1 infection
* No active uncontrolled infection
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* Recovered from prior intensive chemotherapy

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08-16 (Actual); Primary Completion 2009-11-11 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pawlowska, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen I (FTBI, Cyclophosphamide, Fludarabine): Patients undergo FTBI 2-3 times a day on days -9 to -6 for a total of 11 fractions. Patients also receive cyclophosphamide IV over 2 hours on days -5 and -4 and fludarabine phosphate IV on days -5 to -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  filgrastim
  Cyclophosphamide
  Cyclosporine
  Fludarabine phosphate
  Mycophenolate Mofetil
  allogeneic hematopoietic stem cell transplantation
  umbilical cord blood transplantation
  Fractionated total body irradiation
- Regimen II (Busulfan, Fludarabine, Melphalan): Patients receive a test dose of busulfan on day -10 and then dose adjusted busulfan IV 3-4 times daily on days -9 to -6, melphalan IV on days -5 and -4, and fludarabine phosphate IV on days -5 to -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  filgrastim
  Busulfan
  Cyclosporine
  Fludarabine phosphate
  Melphalan
  Mycophenolate Mofetil
  allogeneic hematopoietic stem cell transplantation
  umbilical cord blood transplantation
- Regimen III (TBI, Cyclophosphamide, Fludarabine): Patients receive fludarabine phosphate IV on days -8 to -4 and cyclophosphamide IV over 2 hours on day -3 and undergo TBI (single dose) on day -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  filgrastim
  Cyclophosphamide
  Cyclosporine
  Fludarabine phosphate
  Mycophenolate Mofetil
  allogeneic hematopoietic stem cell transplantation
  umbilical cord blood transplantation
  total-body irradiation
- Regimen IV (Fludarabine, Melphalan): Patients receive fludarabine phosphate IV on days -7 to -3 and melphalan IV on day -2. UCB transplantation: Patients receive 2 combined units of UCB IV on day 0. Patients also receive G-CSF IV or subcutaneously beginning on day 5 (or later) and continuing until blood counts recover. GVHD prophylaxis: Patients receive cyclosporine IV twice daily beginning on day -1 followed by a taper according to institutional guidelines. Patients also receive mycophenolate mofetil orally or IV beginning on day 0 and continuing until day 27 (or as clinically indicated).
  filgrastim
  Cyclosporine
  Fludarabine phosphate
  Melphalan
  Mycophenolate Mofetil
  allogeneic hematopoietic stem cell transplantation
  umbilical cord blood transplantation
- Unassigned: Patients consented but were not eligible for the treatment after screening.
Period: Overall Study
Arm/Group | Regimen I (FTBI, Cyclophosphamide, Fludarabine) | Regimen II (Busulfan, Fludarabine, Melphalan) | Regimen III (TBI, Cyclophosphamide, Fludarabine) | Regimen IV (Fludarabine, Melphalan) | Unassigned
Started | 5 | 0 | 1 | 2 | 2
Completed | 5 | 0 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subject in Regimen II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen I (FTBI, Cyclophosphamide, Fludarabine) | Regimen II (Busulfan, Fludarabine, Melphalan) | Regimen III (TBI, Cyclophosphamide, Fludarabine) | Regimen IV (Fludarabine, Melphalan) | Unassigned | Total
Number analyzed (Participants) | 5 | 0 | 1 | 2 | 2 | 10
Age, Continuous [Median (Full Range); unit: years] | 14 [11 to 18] |  | 58 [58 to 58] | 35 [16 to 54] | 18.5 [9 to 28] | 15 [9 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1 | 1 | 0 | 3
  Male | 4 |  | 0 | 1 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0 | 0 | 0
  Asian | 1 |  | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0 | 0 | 0
  Black or African American | 1 |  | 0 | 0 | 1 | 2
  White | 3 |  | 0 | 2 | 1 | 6
  More than one race | 0 |  | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 1 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at Day 100 After Allogeneic Transplant From Umbilical Cord Blood (UCB)
Description: Number of surviving patients at Day 100 post-transplant divided by number of patients undergone transplantation.
Time Frame: From transplant to Day 100 post-transplant
Population: No subject in the Regimen II arm.
Measure: Number; unit: percentage of surviving patients
Arm/Group | Regimen I (FTBI, Cyclophosphamide, Fludarabine) | Regimen II (Busulfan, Fludarabine, Melphalan) | Regimen III (TBI, Cyclophosphamide, Fludarabine) | Regimen IV (Fludarabine, Melphalan)
Number analyzed (Participants) | 5 | 0 | 1 | 2
percentage of surviving patients | 100 |  | 100 | 100

2. Secondary Outcome: Survival Rate at Day 180 After Allogeneic Transplant From Umbilical Cord Blood (UCB)
Description: Number of surviving patients at Day 180 post-transplant divided by number of patients undergone transplantation.
Time Frame: From transplant up to Day 180 post-transplant
Population: No subject in the Regimen II arm.
Measure: Number; unit: percentage of surviving patients
Arm/Group | Regimen I (FTBI, Cyclophosphamide, Fludarabine) | Regimen II (Busulfan, Fludarabine, Melphalan) | Regimen III (TBI, Cyclophosphamide, Fludarabine) | Regimen IV (Fludarabine, Melphalan)
Number analyzed (Participants) | 5 | 0 | 1 | 2
percentage of surviving patients | 60 |  | 100 | 50

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 100 days post-transplant. All-Cause Mortality monitored/assessed up to 9 years post-transplant.
Description: No subject in the Regimen II arm.
Arm/Group | Regimen I (FTBI, Cyclophosphamide, Fludarabine) | Regimen II (Busulfan, Fludarabine, Melphalan) | Regimen III (TBI, Cyclophosphamide, Fludarabine) | Regimen IV (Fludarabine, Melphalan)
All-Cause Mortality (participants affected / at risk) | 3/5 | 0/0 | 1/1 | 2/2
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/0 | 1/1 | 1/2
Other Adverse Events (participants affected / at risk) | 3/5 | 0/0 | 1/1 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I (FTBI, Cyclophosphamide, Fludarabine) (N=5) | Regimen II (Busulfan, Fludarabine, Melphalan) (N=0) | Regimen III (TBI, Cyclophosphamide, Fludarabine) (N=1) | Regimen IV (Fludarabine, Melphalan) (N=2)
Hemorrhage, GU (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I (FTBI, Cyclophosphamide, Fludarabine) (N=5) | Regimen II (Busulfan, Fludarabine, Melphalan) (N=0) | Regimen III (TBI, Cyclophosphamide, Fludarabine) (N=1) | Regimen IV (Fludarabine, Melphalan) (N=2)
Coagulation - Other (Specify, __) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema:limb (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GU (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (6) | 0 (0) | 1 (1) | 1 (1)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Weight loss (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, __) (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection, Bacterial (COH) (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Infection, Fungal (COH) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, Viral (COH) (Infections and infestations) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Calcium, serum-low (hypocalcemia) (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood alteration (Nervous system disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes